CLINICAL TRIAL: NCT05049486
Title: Computational Model of SNS Using Tractography
Brief Title: Computational Model of SNS (Sacral Nerve Stimulation) Induced Electrical Current Flow Using Tractography Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: London North West NHS Trust
Record Dates: First submitted 2018-04-16; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2018-04

CONDITIONS: Faecal Incontinence
Keywords: Sacral Nerve Stimulator;; DTI;; MRI;; Faecal Incontinence;; CT scan;
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI sequences and (DTI) (No Intervention): The aim of this study is to obtain finer details of tissues surrounding a lead in the pelvis using a combination of high resolution anatomical MRI sequences and diffusion tensor imaging (DTI). To do so, the patient will undergo a MRI scan (3 Tesla) of the pelvis using sequences including anatomical sequences and diffusion tensor imaging technique for construction of sacral nerve tractography prior to permanent SNS. This will be performed over an hour: first 30 minutes for anatomical sequences and the second 30 minutes for DTI sequencing.
- CT scan (Active Comparator): Three to 4 weeks after the procedure the patient will undergo a limited CT scan of the pelvis to visualise the position of the SNS lead. The scan will focus only on the sacrum, implanted lead, and rectum and will not be extended beyond this area. Imaging from this CT will be superimposed to the MRI imaging the patient had pre-operatively, and a computational simulation will be performed.
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — Patients will undergone a pelvic CT scan.
  Arms: CT scan

SUMMARY:
This study aims to obtain finer details of tissues surrounding a lead in the pelvis using a combination of high-resolution anatomical MRI sequences and diffusion tensor imaging (DTI). DTI is a non-invasive technique sometimes described as fiber tractography that enables visualization of the pathways and integrity of nerves. In this feasibility study, we plan to use DTI to assess the sacral plexus and its peripheral nerves. A model will be constructed by superimposing SNS lead from a CT scan onto the DTI imaging to map out the electrode position. It is hoped that this study will lead to a better understanding of both therapeutic and adverse stimulation effects and enable patient-specific adjustments of stimulation parameters.

DETAILED DESCRIPTION:
Patients who have had successful temporary SNS and awaiting permanent SNS will be approached. An assessment will be made to determine whether the patient meets the inclusion/exclusion criteria. Patients will be given a consent form to sign.

The investigators will recruit from the outpatient clinic a total of ten patients for this study.

A physical examination will be performed as per standard practice. Patients will be asked to fill in questionnaires probing the severity of faecal incontinence symptoms. Included questionnaires are ICIQ-B4, Wexner's and St Mark's.

Incontinence score (see appendix). It will also evaluate any existing pain symptoms.

The patient will undergo an MRI scan (3 Tesla) of the pelvis using sequences including anatomical sequences and diffusion tensor imaging technique for construction of sacral nerve tractography prior to permanent SNS. This will be performed at Mount Vernon Hospital over an hour: first 30 minutes for anatomical sequences and the second 30 minutes for DTI sequencing.

A surgical procedure (implant of SNS) will be performed as per standard practice.

Briefly, an antibiotic will be given at induction of anesthesia prior to skin incision. All types of equipment for SNS implantation will be soaked in antibiotic solution (gentamicin 80mg in 500ml of normal saline or equivalent). Under general anesthesia without neuromuscular junction blockade and the patient in prone position, a permanent quadripolar lead (model 3889) will be inserted aiming to observe contraction of the anus and/or toe flexion, which are signs to confirm that the lead is nearby third sacral nerve root. The lead position will be confirmed by an x-ray and the lead will be connected to an implantable neurostimulator which will be placed under the skin but deep enough in the upper outer area of the buttock region. The procedure will be performed according to the manufacturer's manual as per our clinical standard.

After the implantation, patients will be given one generic starting program to start the therapy.

Three to 4 weeks after the procedure the patient will undergo a limited CT scan of the pelvis to visualise the position of the SNS lead. The scan will focus only on the sacrum, implanted lead, and rectum and will not be extended beyond this area. Imaging from this CT will be superimposed to the MRI imaging the patient had pre-operatively, and a computational simulation will be performed (see details below).

After the scan, a clinician will test stimulation settings systematically to find an optimal program. Briefly, as the lead as 4 electrodes, each electrode will be tested, followed by a combination of electrodes. The patient's subjective responses (type and site of sensation, if there is any pain/discomfort site and nature, a degree of pain using a Lickert scale,) will be recorded. The investigators will try and obtain motor response if possible, at the level when patients' anus contracts slightly if this is achievable without causing significant distress and pain to the patients. This is also a routine process and the clinician will note if there is any specific setting that causes adverse pain and identify settings that are comfortable and give stimulation sensation around the anus.

The computational model will be done in a computer laboratory and the record will be compared and evaluated for any clinical relevance. The same set of questionnaires used during the baseline evaluation will be repeated at follow-ups, as per routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are psychologically stable and suitable for intervention and able to provide informed consent
* Patients with symptoms of faecal incontinence for solid or liquid stool
* Patients who have had successful outcome from temporary SNS
* Patients who are willing and competent to fill in questionnaires and undergo an extra CT and MRI scan during the study

Exclusion Criteria:

* Patients who are claustrophobic to undertake MRI scan
* Patients who had previous devices implanted that may be magnetically, electrically, mechanically activated or affected by MRI scan
* Pregnant patients
* Patients who are breastfeeding
* Patients who are psychologically unstable and unsuitable for intervention and unable to provide informed consent
* Patients who did not successfully pass the trial of SNS temporary SNS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Implanting a lead around a nerve for finer details of tissues surrounding a sacral nerve stimulation lead. | 12 months
  Size and distance of the sacral nerves from the implanted lead measured in millimetres (mm).

SECONDARY OUTCOMES:
Stimulation of the sacral nerve using computational model induced electrical current to establish therapeutic range of SNS | 12 months
  Patient's sensation of stimulation will be measured in amplitude (reported in voltage) shown in the standard remote control during the patient stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Carolynne Vaizey, FRCS, Principal Investigator — London North West NHS Trust
Locations (1):
- London North West NHS Trust, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD. Reserach results will be shared at the end of the study by local conferences and by peer scientific journals.

REFERENCES:
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Result] Maeda Y, Lundby L, Buntzen S, Laurberg S. Outcome of sacral nerve stimulation for fecal incontinence at 5 years. Ann Surg. 2014 Jun;259(6):1126-31. doi: 10.1097/SLA.0b013e31829d3969. PMID 23817505
- [Result] Maeda Y, Lundby L, Buntzen S, Laurberg S. Suboptimal outcome following sacral nerve stimulation for faecal incontinence. Br J Surg. 2011 Jan;98(1):140-7. doi: 10.1002/bjs.7302. Epub 2010 Oct 27. PMID 21136568
- [Result] van der Jagt PK, Dik P, Froeling M, Kwee TC, Nievelstein RA, ten Haken B, Leemans A. Architectural configuration and microstructural properties of the sacral plexus: a diffusion tensor MRI and fiber tractography study. Neuroimage. 2012 Sep;62(3):1792-9. doi: 10.1016/j.neuroimage.2012.06.001. Epub 2012 Jun 13. PMID 22705377
- [Result] Cotterill N, Norton C, Avery KN, Abrams P, Donovan JL. A patient-centered approach to developing a comprehensive symptom and quality of life assessment of anal incontinence. Dis Colon Rectum. 2008 Jan;51(1):82-7. doi: 10.1007/s10350-007-9069-3. Epub 2007 Nov 15. PMID 18008106